CLINICAL TRIAL: NCT05549869
Title: Assessment of Serum Leptin in Vitiligo Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Zaghloul Amin, dermatology and andrology resident in luxor international hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-22-09-02
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Active Comparator): obese with vitligo
  Interventions: Diagnostic Test: serum leptin
- group b (Active Comparator): obese without vitligo
  Interventions: Diagnostic Test: serum leptin
- group C (Active Comparator): non obese with vitiligo
  Interventions: Diagnostic Test: serum leptin
- group D (Active Comparator): non obese without vitiligo
  Interventions: Diagnostic Test: serum leptin

INTERVENTIONS:
Diagnostic Test: serum leptin — Evaluation of serum leptin in vitiligo patients and control Assessing its correlation to the body mass index leptin is supposed to contribute to vitiligo pathogenesis through promoting the release of pro-inflammatory mediators

SUMMARY:
Evaluation of serum leptin in vitiligo patients and control Assessing its correlation to the body mass index and disease dermographic data .

DETAILED DESCRIPTION:
, leptin is supposed to contribute to vitiligo pathogenesis through promoting the release of pro-inflammatory mediators such as tumor necrosis factor α "TNF," IL-2 and IL-6, as well as enhancing cytotoxic T cells "CD8" recruitment and inhibiting the functions of regulatory T cells "Tregs". Leptin can also aid in induction of oxidative stress by activating nicotinamide adenine dinucleotide phosphate (NADPH) oxidase• Venous blood samples will be taken from patients and controls to evaluate serum leptin: Morning samples will be taken after 12-h overnight fast in plain vacutainer tubes and directly centrifuged (1098 g for 15 min).

* Sera will be then collected in plain, capped, 5 ml centrifuge tubes "Eppendorf" and freezed at -20ᵒC in a well-monitored freezer until the analysis is performed• Serum leptin will be quantitatively assessed in vitro using DRG leptin Sandwich Enzyme Linked Immuno-Sorbent Assay "ELISA".
* ELISA will be performed according to manufacturer's guidelines where each run included a standard curve.
* Using the mean absorbance value for each sample, the corresponding concentration from the standard curve will be determined.

ELIGIBILITY:
Inclusion Criteria:

* All patients with vitiligo who are above the age of 18 years

Exclusion Criteria:

* Patients with other autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
level of serum leptin | 6 month
  Evaluation of serum leptin in vitiligo patients and control Assessing its correlation to the body mass index and disease dermographic data .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bergqvist C, Ezzedine K. Vitiligo: A Review. Dermatology. 2020;236(6):571-592. doi: 10.1159/000506103. Epub 2020 Mar 10. PMID 32155629
- [Background] Schneider BJ, Naidoo J, Santomasso BD, Lacchetti C, Adkins S, Anadkat M, Atkins MB, Brassil KJ, Caterino JM, Chau I, Davies MJ, Ernstoff MS, Fecher L, Ghosh M, Jaiyesimi I, Mammen JS, Naing A, Nastoupil LJ, Phillips T, Porter LD, Reichner CA, Seigel C, Song JM, Spira A, Suarez-Almazor M, Swami U, Thompson JA, Vikas P, Wang Y, Weber JS, Funchain P, Bollin K. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: ASCO Guideline Update. J Clin Oncol. 2021 Dec 20;39(36):4073-4126. doi: 10.1200/JCO.21.01440. Epub 2021 Nov 1. PMID 34724392
- [Background] Aryanian Z, Shirzadian A, Farzaneh S, Goodarzi A, Azizpour A, Hatami P. Metabolic derangement in patients with vitiligo: a cross-sectional study. J Investig Med. 2022 Apr;70(4):963-966. doi: 10.1136/jim-2021-002062. Epub 2022 Feb 15. PMID 35169000
- [Background] de Oliveira Dos Santos AR, de Oliveira Zanuso B, Miola VFB, Barbalho SM, Santos Bueno PC, Flato UAP, Detregiachi CRP, Buchaim DV, Buchaim RL, Tofano RJ, Mendes CG, Tofano VAC, Dos Santos Haber JF. Adipokines, Myokines, and Hepatokines: Crosstalk and Metabolic Repercussions. Int J Mol Sci. 2021 Mar 5;22(5):2639. doi: 10.3390/ijms22052639. PMID 33807959
- [Background] Mechanick JI, Zhao S, Garvey WT. Leptin, An Adipokine With Central Importance in the Global Obesity Problem. Glob Heart. 2018 Jun;13(2):113-127. doi: 10.1016/j.gheart.2017.10.003. Epub 2017 Dec 13. PMID 29248361